CLINICAL TRIAL: NCT02263209
Title: Prospective Clinical Investigation to Determine the Safety of Taperloc Stems With BioGuard Coating and Exceed ABT Taperfit Acetabular Cups With BioGuard Coating When Used in Cementless Total Hip Arthroplasty
Brief Title: Investigation to Determine Safety of Taperloc Stems With BioGuard Coating When Used in Cementless Total Hip Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU77
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioguard Group (Experimental): Randomised study to either Bioguard or control stock
  Interventions: Device: Bioguard Group
- Control Group (Active Comparator): Randomised study to either Bioguard or control stock
  Interventions: Device: Control Group

INTERVENTIONS:
Device: Bioguard Group — Patients randomised to receive the study investigative device will receive a Bioguard implant
  Other Names: Bioguard device
  Arms: Bioguard Group
Device: Control Group — Patients randomised to receive the control device will receive a Exceed Taperlock implant
  Other Names: Exceed Taperlock
  Arms: Control Group

SUMMARY:
Prospective clinical investigation to determine the safety of Taperloc stems with BioGuard coating and Exceed ABT Taperfit acetabular cups with BioGuard coating when used in cementless total hip arthroplasty

DETAILED DESCRIPTION:
Bioguard Safety Study: Prospective clinical investigation to determine the safety of Taperloc stems with BioGuard coating and Exceed ABT Taperfit acetabular cups with BioGuard coating when used in cementless total hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Eligible for cementless primary total hip arthroplasty according to the Surgical Technique brochure (Appendix 10): "The Taperloc Porous Primary Hip and Exceed ABT Taperfit Prostheses are marketed for non-cemented use in skeletally mature patients undergoing primary hip replacement surgery of non inflammatory degenerative joint disease."
* Under 80 and over 40 years of age
* A pre-operative level of pain and function the same as for conventional joint replacement.
* A likelihood of obtaining relief of pain and improved function
* Full skeletal maturity
* Ability to follow instructions
* Good general health for age
* Willing to return for follow-up evaluations

Exclusion Criteria:

* Patients aged over 80 and under 40 years
* Known allergy to any antibiotics
* Active infection
* Revision arthroplasty
* Marked bone loss which could preclude or compromise adequate fixation of the device
* Uncooperative subjects
* Parkinson's Disease
* Vascular insufficiency of the affected limb, which could compromise bony ingrowth/implant fixation, i.e., diabetes.
* Severe instability or deformity of the ligaments and/or surrounding soft tissue which may preclude stability of the device
* Pregnancy
* BMI > 40
* Use of immunosuppressive drugs
* Women of child bearing potential

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in normalised peri-implant BMD as measured by DXA | 6 months post operative

CONTACTS AND LOCATIONS:
Overall Officials: Sudheer Karlakki, MD, Principal Investigator — RJAH, Oswestry
Locations (1):
- RJAH, Oswestry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided